CLINICAL TRIAL: NCT04693156
Title: Comparison of the Analgesic Effects of Oblique Subcostal, Posterior or Dual Transversus Abdominis Plane (TAP) Block in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Comparison of Oblique Subcostal, Posterior or Dual Transversus Abdominis Plane Block in Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ceylan Saygili (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Sponsor-Investigator, Ceylan Saygili, Resident Doctor, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 132002
Record Dates: First submitted 2020-12-25; First posted 2021-01-05 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Laparoscopic Cholecystectomy; Cholelithiasis; Postoperative Analgesia
Keywords: Transversus Abdominis Plane Block
MeSH Terms: conditions — Cholelithiasis | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- oblique subcostal tap block (Active Comparator): ultrasound-guided right oblique subcostal TAP block with an anesthetic solution of %0.5 Bupivacaine 10ml + %1 Prilocaine 10ml + %0.9 NaCl (sodium chloride) 10ml and ultrasound-guided posterior TAP block with %0.9 NaCl 30ml
  Interventions: Procedure: unilateral ultrasound-guided oblique subcostal TAP block with %0.5 Bupivacaine 10ml + %1 Prilocaine 10ml + %0.9 NaCl 10ml; Procedure: unilateral ultrasound-guided posterior TAP block with %0.9 NaCl 30ml
- posterior tap block (Active Comparator): ultrasound-guided right oblique subcostal TAP block with %0.9 NaCl 30ml and ultrasound-guided posterior TAP block with an anesthetic solution of %0.5 Bupivacaine 10ml + %1 Prilocaine 10ml + %0.9 NaCl 10ml
  Interventions: Procedure: unilateral ultrasound-guided oblique subcostal TAP block with %0.9 NaCl 30ml; Procedure: unilateral ultrasound-guided posterior TAP block with %0.5 Bupivacaine 10ml + %1 Prilocaine 10ml + %0.9 NaCl 10ml
- dual tap block (Active Comparator): ultrasound-guided right oblique subcostal TAP block with %0.5 Bupivacaine 10ml + %1 Prilocaine 10ml + %0.9 NaCl 10ml and ultrasound-guided posterior TAP block with an anesthetic solution of %0.5 Bupivacaine 10ml + %1 Prilocaine 10ml + %0.9 NaCl 10ml
  Interventions: Procedure: unilateral ultrasound-guided oblique subcostal TAP block with %0.5 Bupivacaine 10ml + %1 Prilocaine 10ml + %0.9 NaCl 10ml; Procedure: unilateral ultrasound-guided posterior TAP block with %0.5 Bupivacaine 10ml + %1 Prilocaine 10ml + %0.9 NaCl 10ml

INTERVENTIONS:
Procedure: unilateral ultrasound-guided oblique subcostal TAP block with %0.5 Bupivacaine 10ml + %1 Prilocaine 10ml + %0.9 NaCl 10ml — In the supine position, after the skin sterilization, ultrasound with a high-frequency linear probe will be placed subcostally and from the xiphoid to the right iliac crest obliquely. The rectus abdominis and underlying transversus abdominis muscles will be identified. The local anesthetic solution (%0.5 Bupivacaine 10ml + %1 Prilocaine 10ml + %0.9 NaCl 10ml) will be injected after negative aspiration to the transversus abdominis plane between the rectus abdominis and transversus abdominis muscles along the oblique subcostal line.
  Arms: dual tap block; oblique subcostal tap block
Procedure: unilateral ultrasound-guided oblique subcostal TAP block with %0.9 NaCl 30ml — In the supine position, after the skin sterilization, ultrasound with a high-frequency linear probe will be placed subcostally and from the xiphoid to the right iliac crest obliquely. %0.9 NaCl 30ml will be injected after negative aspiration to the transversus abdominis plane between the rectus abdominis and transversus abdominis muscles along the oblique subcostal line.
  Arms: posterior tap block
Procedure: unilateral ultrasound-guided posterior TAP block with %0.5 Bupivacaine 10ml + %1 Prilocaine 10ml + %0.9 NaCl 10ml — After the oblique subcostal TAP block, the operation table will be slightly turned left laterally for better visualization of the blocking area. The same high-frequency linear ultrasound (Esaote MyLab5) probe will be placed over the postero-lateral abdominal wall, posterior of the mid-axillary line between the costal margin and iliac crest. After the identification of the internal abdominis, transversus abdominis, and quadratus lumborum muscles, the needle will be advanced into the transversus abdominis plane between the internal abdominis and transversus abdominis muscles, at the aponeurosis of quadratus lumborum and these muscles. The local anesthetic solution (%0.5 Bupivacaine 10ml + %1 Prilocaine 10ml + %0.9 NaCl 10ml) will be injected after negative aspiration.
  Arms: dual tap block; posterior tap block
Procedure: unilateral ultrasound-guided posterior TAP block with %0.9 NaCl 30ml — After the oblique subcostal TAP block, the operation table will be slightly turned left laterally for better visualization of the blocking area. The same high-frequency linear ultrasound probe will be placed over the postero-lateral abdominal wall, posterior of the mid-axillary line between the costal margin and iliac crest. After the identification of the internal abdominis, transversus abdominis, and quadratus lumborum muscles, the needle will be advanced into the transversus abdominis plane between the internal abdominis and transversus abdominis muscles, at the aponeurosis of quadratus lumborum and these muscles. %0.9 NaCl 30ml will be injected after negative aspiration.
  Arms: oblique subcostal tap block

SUMMARY:
The aim of the study is to evaluate the difference of postoperative analgesic effects and opioid consumption between ultrasound-guided unilateral oblique subcostal, posterior, or dual TAP blocks in patients undergoing laparoscopic cholecystectomy for cholelithiasis.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy is one of the most frequent operations. Laparoscopic cholecystectomy is a less invasive technic that provides early mobilization and reduces hospitalization time thus preferred to laparotomy often. There is a minimum of 4 trochar incisions on the right side of the abdomen at epigastric, umbilical, midclavicular subcostal, and anterior axillary subcostal regions in laparoscopic cholecystectomy. Some patients have a drainage tube at the middle/lower right abdomen. Thus the right side of the abdomen is the target side for abdominal wall blocks.

Most patients complain of moderate pain after surgery which requiring opioids, mostly in the upper abdomen, lower abdomen, and shoulder. The pain has three components; somatic pain at the anterior abdominal wall, visceral pain caused by pneumoperitoneum and referred shoulder pain. Preventing postoperative pain is important for reducing respiratory complications and hospitalization time also improve patient satisfaction. Opioids are preferred less due to their side effects like nausea-vomiting and respiratory depression although which is preferable for moderate and severe pain. Transversus abdominis plane (TAP) block is the most preferred abdominal wall block to provide effective postoperative pain control for reducing perioperative analgesic requirements like opioids.

TAP block was first described by Rafi by anatomic landmark technic then by Hebbard with ultrasonographic guidance. TAP block is a regional technic and a plan block that blocks the thoracolumbar nerves that innervate the anterior and lateral abdominal wall and passes in between the muscles' internal oblique and transversus abdominis. External oblique, internal oblique, and transversus abdominis muscles are displayed sequentially by ultrasonography. A hypoechoic, spindle-shaped separation of the fascia by hydrodissection technic is performed by local anesthetic injection in between the internal oblique muscle (or rectus abdominis) and transversus abdominis muscle. Dermatomal spread is differentiated with subcostal, oblique subcostal, and posterior approaches.

In oblique subcostal TAP block, anesthetic solution spreads across the location of T6-L1 nerves thus suitable for surgeries at both superior and inferior the umbilicus. Some other studies show that posterior TAP block can block the T5 to L1 thoracolumbar nerves thereby spreading into paravertebral space. The paravertebral spread of the posterior TAP block suggests that the analgesic efficacy will be long-lasting by blocking the thoracolumbar sympathetic chain and will spread to a wider dermatomal area. In this study, the investigators aimed to compare the analgesic efficacy and opioid-sparing effects of oblique subcostal, posterior, and dual TAP blocks in patients undergoing laparoscopic cholecystectomy. Taking the advantage of the paravertebral extension of the posterior approach and the wide spread of the oblique subcostal approach on the anterior abdominal wall, it's supposed to be the dual TAP block will result in lower pain scores.

All patients will have general anesthesia. For premedication midazolam 0.03mg/kg will be used for all patients. At the induction of the anesthesia, patients will receive propofol 2 mg/ kg, fentanyl 2 μg/kg, and rocuronium 0.6 mg/ kg IV. After enough muscle relaxation patients will be orotracheally intubated. General anesthesia will be maintained with sevoflurane and air/O2 mixture. The end-tidal carbon dioxide partial pressure will be maintained between 32 and 36 mmHg by adjusting the pressure-controlled mechanical ventilation. All patients will receive tramadol 1mg/kg, paracetamol 1gr, and ondansetron 8mg intravenously before skin closure. Postoperatively ultrasound-guided right oblique subcostal and posterior TAP blocks will be performed on all patients. Postoperatively starting from at the postoperative care unit (0th hour) then 2nd,4th, 6th, 8th, 12th and 24th hours pain intensity by numerical rating scale (NRS) at rest and with motion, sensory dermatomal involvement by pinprick test, Ramsey sedation scales, nausea and vomiting scores, and rescue analgesic medication requirements will be recorded. Besides heart rate, blood pressure, respiratory rate, peripheric oxygen saturation, mobilization time, side effects if there are any will be recorded at the aforementioned hours. Patients with NRS≥4 will receive dexketoprofen 50mg as rescue analgesic medication. If NRS≥7 tramadol 100mg will be administered.

The study will start after getting written informed consent from patients who are informed about the study and potential risks. The study is a prospective, clinical, randomized controlled, quadruple-blinded, and monocenter study. Participation of the 60 patients undergoing laparoscopic cholecystectomy had been planned. Patients will be randomized into three groups of 20 patients each.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective laparoscopic cholecystectomy for cholelithiasis
* ASA (American Society of Anesthesiologists) I-II

Exclusion Criteria:

* Patient refusal
* Perforation of the gallbladder
* Patients with acute cholecystitis
* History of the previous gallbladder surgery
* Pregnancy
* Morbid obesity
* Psychiatric disorder
* Epilepsia
* Renal insufficiency
* Coagulopathy
* Patients known allergic to drugs used for study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
postoperative pain intensity at rest and with motion | postoperative 0 hour
  postoperative 0th hour Numerical Rating Scale measured on 0-10 ( 0= no pain, 10= the worst imaginable pain) when patient is awake in postanesthesia care unit. This outcome is compared between all three groups.
postoperative pain intensity at rest and with motion | postoperative 2 hours
  postoperative 2nd hour Numerical Rating Scale measured on 0-10 ( 0= no pain, 10= the worst imaginable pain) when patient is on the ward. This outcome is compared between all three groups.
postoperative pain intensity at rest and with motion | postoperative 4 hours
  postoperative 4th hour Numerical Rating Scale measured on 0-10 ( 0= no pain, 10= the worst imaginable pain) when patient is on the ward. This outcome is compared between all three groups.
postoperative pain intensity at rest and with motion | postoperative 6 hours
  postoperative 6th hour Numerical Rating Scale measured on 0-10 ( 0= no pain, 10= the worst imaginable pain) when patient is on the ward. This outcome is compared between all three groups.
postoperative pain intensity at rest and with motion | postoperative 8 hours
  postoperative 8th hour Numerical Rating Scale measured on 0-10 ( 0= no pain, 10= the worst imaginable pain) when patient is on the ward. This outcome is compared between all three groups.
postoperative pain intensity at rest and with motion | postoperative 12 hours
  postoperative 12th hour Numerical Rating Scale measured on 0-10 ( 0= no pain, 10= the worst imaginable pain) when patient is on the ward. This outcome is compared between all three groups.
postoperative pain intensity at rest and with motion | postoperative 24 hours
  postoperative 24th hour Numerical Rating Scale measured on 0-10 ( 0= no pain, 10= the worst imaginable pain) when patient is on the ward. This outcome is compared between all three groups.

SECONDARY OUTCOMES:
postoperative opioid consumption | 24 hours
  opioids given at post-anaesthesia care unit and ward
postoperative dermatomal level of sensory block | 24 hours
  postoperative 0.,2.,4.,6.,8.,12. and 24.hours via pinprick test
postoperative sedation | 24 hours
  postoperative 0.,2.,4.,6.,8.,12. and 24.hours Ramsey Sedation Scale; (1) anxious and agitated or restless or both; (2) co-operative, oriented and tranquil; (3) responding to commands only; (4) brisk response to light glabellar tap or loud auditory stimulus; (5) sluggish response to light glabellar tap or loud auditory stimulus; (6) no response to stimulus.
postoperative nausea and vomiting | 24 hours
  postoperative 0.,2.,4.,6.,8.,12. and 24.hours Nausea and Vomiting Score; (0) without nausea or vomiting; (1) nausea without vomiting; (2) one episode of vomiting; (3) two or more episode of vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Fatis Altındas, Prof. Dr., Study Director — Istanbul University-Cerrahpasa, Cerrahpasa Medical Faculty, Anesthesiology and Reanimation; Emre S Erbabacan, Asc.Prof, Study Chair — Istanbul University-Cerrahpasa, Cerrahpasa Medical Faculty, Anesthesiology and Reanimation; Aylin Ozdilek, Asc.Prof, Study Chair — Istanbul University-Cerrahpasa, Cerrahpasa Medical Faculty, Anesthesiology and Reanimation; Cigdem Akyol Beyoglu, M.D., Study Chair — Istanbul University-Cerrahpasa, Cerrahpasa Medical Faculty, Anesthesiology and Reanimation; Ceylan Saygili, M.D., Principal Investigator — Istanbul University-Cerrahpasa, Cerrahpasa Medical Faculty, Anesthesiology and Reanimation
Locations (1):
- Cerrahpasa Medical Faculty General Surgery Operating Theater, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD (individual participant data) available to other researchers

REFERENCES:
- [Background] Ure BM, Troidl H, Spangenberger W, Dietrich A, Lefering R, Neugebauer E. Pain after laparoscopic cholecystectomy. Intensity and localization of pain and analysis of predictors in preoperative symptoms and intraoperative events. Surg Endosc. 1994 Feb;8(2):90-6. doi: 10.1007/BF00316616. PMID 8165491
- [Background] Alexander JI. Pain after laparoscopy. Br J Anaesth. 1997 Sep;79(3):369-78. doi: 10.1093/bja/79.3.369. No abstract available. PMID 9389858
- [Background] Wills VL, Hunt DR. Pain after laparoscopic cholecystectomy. Br J Surg. 2000 Mar;87(3):273-84. doi: 10.1046/j.1365-2168.2000.01374.x. PMID 10718794
- [Background] Rafi AN. Abdominal field block: a new approach via the lumbar triangle. Anaesthesia. 2001 Oct;56(10):1024-6. doi: 10.1046/j.1365-2044.2001.02279-40.x. No abstract available. PMID 11576144
- [Background] Tsai HC, Yoshida T, Chuang TY, Yang SF, Chang CC, Yao HY, Tai YT, Lin JA, Chen KY. Transversus Abdominis Plane Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:8284363. doi: 10.1155/2017/8284363. Epub 2017 Oct 31. PMID 29226150
- [Background] Hebbard P, Fujiwara Y, Shibata Y, Royse C. Ultrasound-guided transversus abdominis plane (TAP) block. Anaesth Intensive Care. 2007 Aug;35(4):616-7. No abstract available. PMID 18020088
- [Background] Jankovic Z, Ahmad N, Ravishankar N, Archer F. Transversus abdominis plane block: how safe is it? Anesth Analg. 2008 Nov;107(5):1758-9. doi: 10.1213/ane.0b013e3181853619. No abstract available. PMID 18931248
- [Background] Hebbard PD, Barrington MJ, Vasey C. Ultrasound-guided continuous oblique subcostal transversus abdominis plane blockade: description of anatomy and clinical technique. Reg Anesth Pain Med. 2010 Sep-Oct;35(5):436-41. doi: 10.1097/aap.0b013e3181e66702. PMID 20830871
- [Background] Carney J, Finnerty O, Rauf J, Bergin D, Laffey JG, Mc Donnell JG. Studies on the spread of local anaesthetic solution in transversus abdominis plane blocks. Anaesthesia. 2011 Nov;66(11):1023-30. doi: 10.1111/j.1365-2044.2011.06855.x. Epub 2011 Aug 18. PMID 21851346
- [Background] Abdallah FW, Laffey JG, Halpern SH, Brull R. Duration of analgesic effectiveness after the posterior and lateral transversus abdominis plane block techniques for transverse lower abdominal incisions: a meta-analysis. Br J Anaesth. 2013 Nov;111(5):721-35. doi: 10.1093/bja/aet214. Epub 2013 Jun 27. PMID 23811424
- [Background] McDonnell JG, O'Donnell BD, Farrell T, Gough N, Tuite D, Power C, Laffey JG. Transversus abdominis plane block: a cadaveric and radiological evaluation. Reg Anesth Pain Med. 2007 Sep-Oct;32(5):399-404. doi: 10.1016/j.rapm.2007.03.011. PMID 17961838
- [Background] Bhatia N, Arora S, Jyotsna W, Kaur G. Comparison of posterior and subcostal approaches to ultrasound-guided transverse abdominis plane block for postoperative analgesia in laparoscopic cholecystectomy. J Clin Anesth. 2014 Jun;26(4):294-9. doi: 10.1016/j.jclinane.2013.11.023. Epub 2014 Jun 2. PMID 24882606
- [Background] Katz J, Melzack R. Measurement of pain. Surg Clin North Am. 1999 Apr;79(2):231-52. doi: 10.1016/s0039-6109(05)70381-9. PMID 10352653